CLINICAL TRIAL: NCT00486135
Title: A Phase 1 Dose-Escalation Study of the Safety and Pharmacokinetics of XL147 Administered Orally Daily to Subjects With Solid Tumors or Lymphoma
Brief Title: Study of the Safety and Pharmacokinetics of XL147 (SAR245408) in Adults With Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TED11433; XL147-001 (Other: Other study code)
Record Dates: First submitted 2007-06-11; First posted 2007-06-13 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Cancer; Lymphoma
Keywords: Cancer; Solid tumors; Lymphoma
MeSH Terms: conditions — Neoplasms; Lymphoma | interventions — XL147

ARMS (3):
- 1 (Experimental): Daily dosing for 21 days/7 days off
  Interventions: Drug: XL147 (SAR245408)
- 2 (Experimental): Continuous daily dosing
  Interventions: Drug: XL147 (SAR245408)
- 3 (Experimental): Continuous daily dosing
  Interventions: Drug: XL147 (SAR245408)

INTERVENTIONS:
Drug: XL147 (SAR245408) — Gelatin capsules supplied in 25-mg and 100-mg dosage strengths
  Arms: 1; 2
Drug: XL147 (SAR245408) — Tablets supplied as 100-mg, 150-mg, and 200-mg dosage strengths
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of XL147 in subjects with solid tumors or lymphoma. Both a capsule and a tablet formulation will be evaluated. XL147 is a new chemical entity that inhibits PI3 Kinase. Inactivation of PI3K has been shown to inhibit growth and induce apoptosis (programmed cell death) in tumor cells.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has a histologically confirmed solid tumor that is metastatic or unresectable, and for which standard curative or palliative measures do not exist or are no longer effective, and there are no known therapies to prolong survival. An expanded cohort will be enrolled; NSCLC subjects enrolled must have a diagnosis of relapsed or refractory NSCLC (Stage IIIB or IV) and have received at least two prior regimens including one platinum-based chemotherapy regimen.
2. The subject has a histologically confirmed diagnosis of lymphoma which is relapsed or refractory to standard therapy.
3. For subjects with solid tumors, the subject has disease that is assessable by tumor marker, physical, or radiologic means. There are separate criteria that apply to subjects with lymphoma.
4. Subjects with indolent lymphoma must have documented disease status within 12 months prior to study entry.
5. The subject is ≥18 years old.
6. The subject's weight is ≥40 kg.
7. The subject has an Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
8. The subject has adequate organ and marrow function, and a fasting plasma glucose (FPG) <160 mg/dL and HbA1c of <8% at screening.
9. For the subjects with solid tumors who are to be enrolled into the expanded MTD cohort and tumor genetic alteration subjects:

   1. tumor tissue amenable to serial biopsy, and
   2. additional informed consent.
10. The subject is capable of understanding and complying with the protocol and has signed the informed consent document.
11. Sexually active subjects (male and female) must use medically acceptable methods of contraception during the course of the study and for 3 months following discontinuation of study drug.
12. Female subjects of childbearing potential must have a negative serum pregnancy test at screening.
13. At least ten 4-10 micron tissue sections, archival or fresh, or a tissue block, of the subject's tumor should be identified and designated for shipment to the sponsor where allowed by local regulatory bodies. For subjects with lymphoma, tissue from an excisional or core biopsy or, in case of marrow involvement, a bone marrow aspirate/biopsy is acceptable.

Exclusion Criteria:

1. The subject has previously been treated with a selective PI3K inhibitor.
2. Additional restrictions on prior treatment apply.
3. For lymphoma subjects: known central nervous system involvement, autoimmune disease requiring immunosuppressive therapy, systemic treatment with prednisone >20mg/day or equivalent within 2 weeks prior to first dose of XL147, autologous stem cell transplantation within 12 weeks prior to first dose, history of any allogeneic transplantation.
4. The subject has not recovered from toxicity due to all prior therapies.
5. The subject has a primary brain tumor. Subjects with brain metastasis are considered eligible if the subject has not received radiation therapy for brain metastasis within 2 weeks of enrollment and has been on a stable dose of steroids for 2 or more weeks.
6. The subject is currently receiving anticoagulation with therapeutic doses of warfarin (low-dose warfarin is permitted).
7. The subject has prothrombin time/partial thromboplastin time (PT/PTT) or International Normalized Ratio (INR) test results at screening that are above 1.3x the laboratory upper limit of normal.
8. The subject has an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
9. The subject has psychiatric illness/social situation(s) that would limit compliance with study requirements.
10. The subject is pregnant or breastfeeding.
11. The subject is known to be positive for the human immunodeficiency virus (HIV).
12. The subject has a previously identified allergy or hypersensitivity to components of the XL147 formulation.
13. The subject has a baseline corrected QT interval (QTc) >460 ms.
14. The subject is unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2007-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Safety, tolerability, and maximum tolerated dose of oral administration of two formulations of XL147 in two treatment schedules | Assessed at each visit/periodic visits
Safety and tolerability of oral dosing with XL147 capsules in subjects with lymphoma, and of XL147 capsules and tablets in subjects with solid tumors | Assessed at periodic study visits

SECONDARY OUTCOMES:
Plasma pharmacokinetics of daily oral administration of XL147 in two treatment schedules | Assessed during periodic visits
Pharmacodynamic effects of XL147 on tumor tissue when administered at the maximum tolerated dose in two treatment schedules | Assessed during periodic visits after MTD is determined
Plasma pharmacokinetics of XL147 capsule and tablet formulations | Assessed during periodic visits after the preliminary MTD for the continuous daily dosing schedule is determined

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (4):
- United States (3):
  - Investigational Site Number 1241, Augusta, Georgia
  - Investigational Site Number 1503, Boston, Massachusetts
  - Investigational Site Number 1401, Dallas, Texas
- Investigational Site Number 3412, Barcelona, Spain

REFERENCES:
- [Derived] Edelman G, Rodon J, Lager J, Castell C, Jiang J, Van Allen EM, Wagle N, Lindeman NI, Sholl LM, Shapiro GI. Phase I Trial of a Tablet Formulation of Pilaralisib, a Pan-Class I PI3K Inhibitor, in Patients with Advanced Solid Tumors. Oncologist. 2018 Apr;23(4):401-e38. doi: 10.1634/theoncologist.2017-0691. Epub 2018 Mar 28. PMID 29593099